CLINICAL TRIAL: NCT04395885
Title: Sexual Function Among Egyptian Healthcare Professionals During COVID 19 Pandemic
Brief Title: Sexual Function During COVID 19 Pandemic
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: SFCOV
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: health care staff, regardless of gender, who is actively working during the outbreak
  Interventions: Other: Electronic questionnaire
- control group: age matched group of non-health worker individuals.
  Interventions: Other: Electronic questionnaire

INTERVENTIONS:
Other: Electronic questionnaire — Assess the current sexuality according to the gender using sexual questionnaires for men and women were adapted from the Arabic validated version of the five-item International Index of Erectile Function which is a validated, multidimensional, self-administered questionnaire used for the clinical assessment of erectile dysfunction.and for female Arabic validated version of the Female Sexual Function Index

SUMMARY:
The outbreak of a new Coronavirus disease (COVID-19), caused by the 2019-nCoV infection in December 2019 is one of the most severe global epidemic health problems.The rapid contagion of this Novel virus has provoked the World Health Organization (WHO) to classifying the outbreak as a "Public Health Emergency of International Concern" on January 30 2020 to a "Pandemic" on March 11th 2020

ELIGIBILITY:
Inclusion Criteria:

* health care staff
* working during the outbreak

Exclusion Criteria:

* refuse to participate

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: health care staff, regardless of gender, who is actively working during the outbreak, will be invited to participate in this study by filling anonyms electronic survey. And an age matched group of non-health worker individuals.
Sampling Method: Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
The percentage of study participants diagnosed with sexual dysfunction | one month
  The diagnosis will be made based on the score results

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ahmed Abbas, Assiut, Cairo Governorate
  - Assiut Faculty of Medicine, Asyut

IPD SHARING:
Plan to Share IPD: No